CLINICAL TRIAL: NCT03740243
Title: Comparison of Buprenorphine vs Buprenorphine/Naloxone on the Effects of Maternal Symptomatology
Brief Title: Buprenorphine vs Buprenorphine/Naloxone on the Effects of Maternal Symptomatology
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, David Garry DO, Director, Maternal Fetal Medicine, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1175806
Record Dates: First submitted 2018-10-15; First posted 2018-11-14 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Opioid-use Disorder
Keywords: opioid use disorder; Buprenorphine/naloxone; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine; Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- buprenorphine (Active Comparator): Buprenorphine 2 mg to 8 mg daily: Light to moderate history of opioid use (heroin, oxycodone, etc.) and/or Clinical Opioid Withdraw Scale (COWS) scores 5-24
  Buprenorphine 8 mg to 16 mg daily: Heavy history of opioid use (heroin, oxycodone, etc.) and/or Clinical Opioid Withdraw Scale (COWS) scores 25-36+
  Interventions: Drug: Buprenorphine
- buprenorphine/naloxone (Experimental): Buprenorphine/naloxone 4 mg/1 mg daily once daily or twice daily (BID): Light to moderate history of opioid use (heroin, oxycodone, etc.) and/or Clinical Opioid Withdraw Scale (COWS) scores 5-24
  Buprenorphine/naloxone 8 mg/2 mg daily once daily or twice daily (BID): Heavy history of opioid use (heroin, oxycodone, etc.) and/or Clinical Opioid Withdraw Scale (COWS) scores 25-36+
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Buprenorphine/naloxone tablet or film
  Other Names: suboxone, bunavail, zubsolv
  Arms: buprenorphine/naloxone
Drug: Buprenorphine — Buprenorphine tablet
  Other Names: subutex, belbuca, butrans,sublocade
  Arms: buprenorphine

SUMMARY:
This study will assesses the efficacy of buprenorphine/naloxone vs buprenorphine on maternal withdrawal symptoms and drug cravings.

This is a randomized controlled trial to a cohort of pregnant women seeking medication-assisted treatment for opioid use disorders. Half of participants will receive buprenorphine, while the other half of participants receive a combination of buprenorphine/naloxone

DETAILED DESCRIPTION:
Buprenorphine and Buprenorphine/naloxone each are used to treat opioid use disorders in pregnancy.

Buprenorphine has many preferential characteristics over methadone including decreased risk of maternal overdose, lower incidence of preterm labor, less frequent clinical visits, shorter duration of neonatal hospital stay and treatment for neonatal abstinence syndrome. Recent studies have found that increasing the dosing frequencies of buprenorphine is more efficacious to prevent maternal withdrawal symptoms, improve compliance, and theoretically produce better pregnancy outcomes.

Buprenorphine/naloxone, a combination opioid of buprenorphine and naloxone, has also been investigated as an alternative to treatment and maintenance for opioid use disorder. The advantage of the combination of buprenorphine with naloxone is that it reduces the potential for abuse. As a partial mu opioid agonist, buprenorphine alone has the capacity to induce typical opioid effects such as euphoria, which are enhanced when the drug is taken intravenously. By combining buprenorphine with naloxone, an opioid antagonist, the capacity for buprenorphine to be abused is reduced.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* With a confirmed viable intrauterine pregnancy
* Opioid Use Disorder
* Care in a Stony Brook Medicine OBGYN clinical office sites
* Medication-assisted treatment through Stony Brook Medicine OBGYN office sites

Exclusion Criteria:

* Known or suspected allergy to buprenorphine or buprenorphine/naloxone
* Carrying a fetus with known aneuploidy or anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — As this study pertains only to pregnant patients seeking treatment for opioid use disorders, females are the only biologically plausiable participants.
Enrollment: 0 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Compliance antepartum | From entry into the study until delivery (through study completion, an average of 9 months which is duration of the pregnancy)
  To compare compliance with buprenorphine versus buprenorphine/naloxone medication-assisted treatment (MAT) in pregnant women. Compliance will include the incidence of urine toxicology testing positive for illicit substances during prenatal care and at the time of admission for delivery.
Compliance postpartum | 2 month period postpartum
  To compare compliance with buprenorphine versus buprenorphine/naloxone medication-assisted treatment (MAT) in the postpartum period. Compliance will include the incidence of urine toxicology testing positive for illicit substances from the time of discharge from the hospital following the delivery over a 2 month period postpartum (postpartum period).
Dosing antepartum | From entry into the study until delivery (through study completion, an average of 9 months which is duration of the pregnancy)
  Evaluate all women for the need a significant dosing change in buprenorphine or buprenorphine/naloxone (>50% increase or decrease) during pregnancy.
Dosing postpartum | 2 month period postpartum
  Evaluate all women for the need a significant dosing change in buprenorphine or buprenorphine/naloxone (>50% increase or decrease) from the hospital following the delivery over a 2 month period postpartum (postpartum period).

SECONDARY OUTCOMES:
Maternal Outcomes Withdraw Scoring | Duration of pregnancy and 2 months of postpartum period
  Prenatal Clinical Opioid Withdraw Scale (COWS) score and drug cravings score (0 to 48 score)
  Score interpretation:
  5-12 = Mild 13-24 = Moderate 25-36 = Moderately Severe More than 36 = Severe Withdrawal
Maternal Outcome Metabolites | At delivery of newborn
  Umbilical cord blood levels of metabolites of buprenorphine (norbuprenorphine, buprenorphine glucuronide, and norbuprenorphine glucuronide) which are obtained from the umbilical cord after delivery of the baby (one time specimen for evaluation)
Placental dysmaturity | At delivery of newborn
  Placental histology (obtained at delivery - pathology specimen)
Neonatal Outcomes | Birth until discharge from hospital (performed during hospitalization of newborn from 0 to 30 days of life)
  Neonatal Abstinence Syndrome (NAS) rate
Neonatal stay | Birth to newborn discharge home (from day 0 through 120 days of life)
  Duration of newborn inpatient hospital stay
Newborn | At birth
  Gestational age at birth (range 23 to 43 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: David J Garry, DO, Principal Investigator — Stony Brook University

IPD SHARING:
Plan to Share IPD: No
In regards to the participants and neonates' health information, care will be taken to ensure privacy. All data and specimens will be coded with a case number and de-identified, and exported to a REDcap application system (secure data file approved by Institutional Review Board). The REDcap application data will be kept on the department's secure, shared institutional, server space.

REFERENCES:
- [Result] Committee Opinion No. 711: Opioid Use and Opioid Use Disorder in Pregnancy. Obstet Gynecol. 2017 Aug;130(2):e81-e94. doi: 10.1097/AOG.0000000000002235. PMID 28742676
- [Result] Bastian JR, Chen H, Zhang H, Rothenberger S, Tarter R, English D, Venkataramanan R, Caritis SN. Dose-adjusted plasma concentrations of sublingual buprenorphine are lower during than after pregnancy. Am J Obstet Gynecol. 2017 Jan;216(1):64.e1-64.e7. doi: 10.1016/j.ajog.2016.09.095. Epub 2016 Sep 26. PMID 27687214
- [Result] Caritis SN, Bastian JR, Zhang H, Kalluri H, English D, England M, Bobby S, Venkataramanan R. An evidence-based recommendation to increase the dosing frequency of buprenorphine during pregnancy. Am J Obstet Gynecol. 2017 Oct;217(4):459.e1-459.e6. doi: 10.1016/j.ajog.2017.06.029. Epub 2017 Jun 29. PMID 28669739
- [Result] Chavan NR, Ashford KB, Wiggins AT, Lofwall MR, Critchfield AS. Buprenorphine for Medication-Assisted Treatment of Opioid Use Disorder in Pregnancy: Relationship to Neonatal Opioid Withdrawal Syndrome. AJP Rep. 2017 Oct;7(4):e215-e222. doi: 10.1055/s-0037-1608783. Epub 2017 Dec 7. PMID 29226017
- [Result] Debelak K, Morrone WR, O'Grady KE, Jones HE. Buprenorphine + naloxone in the treatment of opioid dependence during pregnancy-initial patient care and outcome data. Am J Addict. 2013 May-Jun;22(3):252-4. doi: 10.1111/j.1521-0391.2012.12005.x. PMID 23617867
- [Result] Geber WF, Schramm LC. Congenital malformations of the central nervous system produced by narcotic analgesics in the hamster. Am J Obstet Gynecol. 1975 Dec 1;123(7):705-13. doi: 10.1016/0002-9378(75)90492-5. PMID 907
- [Result] Fudala PJ, Bridge TP, Herbert S, Williford WO, Chiang CN, Jones K, Collins J, Raisch D, Casadonte P, Goldsmith RJ, Ling W, Malkerneker U, McNicholas L, Renner J, Stine S, Tusel D; Buprenorphine/Naloxone Collaborative Study Group. Office-based treatment of opiate addiction with a sublingual-tablet formulation of buprenorphine and naloxone. N Engl J Med. 2003 Sep 4;349(10):949-58. doi: 10.1056/NEJMoa022164. PMID 12954743
- [Result] Jumah NA, Edwards C, Balfour-Boehm J, Loewen K, Dooley J, Gerber Finn L, Kelly L. Observational study of the safety of buprenorphine+naloxone in pregnancy in a rural and remote population. BMJ Open. 2016 Oct 31;6(10):e011774. doi: 10.1136/bmjopen-2016-011774. PMID 27799240
- [Result] Lund IO, Fischer G, Welle-Strand GK, O'Grady KE, Debelak K, Morrone WR, Jones HE. A Comparison of Buprenorphine + Naloxone to Buprenorphine and Methadone in the Treatment of Opioid Dependence during Pregnancy: Maternal and Neonatal Outcomes. Subst Abuse. 2013;7:61-74. doi: 10.4137/SART.S10955. Epub 2013 Mar 14. PMID 23531704
- [Result] Mendelson J, Jones RT. Clinical and pharmacological evaluation of buprenorphine and naloxone combinations: why the 4:1 ratio for treatment? Drug Alcohol Depend. 2003 May 21;70(2 Suppl):S29-37. doi: 10.1016/s0376-8716(03)00057-7. PMID 12738348
- [Result] Nguyen L, Lander LR, O'Grady KE, Marshalek PJ, Schmidt A, Kelly AK, Jones HE. Treating women with opioid use disorder during pregnancy in Appalachia: Initial neonatal outcomes following buprenorphine + naloxone exposure. Am J Addict. 2018 Mar;27(2):92-96. doi: 10.1111/ajad.12687. Epub 2018 Feb 23. PMID 29473258
- [Result] Poon S, Pupco A, Koren G, Bozzo P. Safety of the newer class of opioid antagonists in pregnancy. Can Fam Physician. 2014 Jul;60(7):631-2, e348-9. PMID 25022635
- [Result] Simojoki K, Vorma H, Alho H. A retrospective evaluation of patients switched from buprenorphine (Subutex) to the buprenorphine/naloxone combination (Suboxone). Subst Abuse Treat Prev Policy. 2008 Jun 17;3:16. doi: 10.1186/1747-597X-3-16. PMID 18559110
- [Result] Strain EC, Harrison JA, Bigelow GE. Induction of opioid-dependent individuals onto buprenorphine and buprenorphine/naloxone soluble-films. Clin Pharmacol Ther. 2011 Mar;89(3):443-9. doi: 10.1038/clpt.2010.352. Epub 2011 Jan 26. PMID 21270789
- [Result] Wiegand SL, Stringer EM, Stuebe AM, Jones H, Seashore C, Thorp J. Buprenorphine and naloxone compared with methadone treatment in pregnancy. Obstet Gynecol. 2015 Feb;125(2):363-368. doi: 10.1097/AOG.0000000000000640. PMID 25569005

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Protocol and SAP (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03740243/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03740243/ICF_001.pdf
  • Study Protocol: COWS questionnaire and Brief Substance Cravings scale (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT03740243/Prot_002.pdf